CLINICAL TRIAL: NCT04570384
Title: Prospective, Randomized, Double-Blind, Placebo-Controlled Phase II Trial of Intravenous L-Citrulline (Turnobi) to Delay and Potentially Prevent the Need for Invasive Mechanical Ventilation for Acute Hypoxemic Respiratory Failure in Patients With COVID-19 (SARS-CoV-2) Illness
Brief Title: Intravenous L-Citrulline Influence on the Need for Invasive Mechanical Ventilation for Acute Hypoxemic Respiratory Failure in Patients With COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asklepion Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIT-COVID19-002-01
Record Dates: First submitted 2020-09-17; First posted 2020-09-30 (Actual); Results first posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-01

CONDITIONS: Acute Hypoxemic Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Citrulline; serum P-component

STUDY DESIGN:
Intervention Model Description: Placebo controlled and Active Drug
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind Clinical Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IV L-Citrulline (Turnobi) Arm (Active Comparator): Patients randomized to citrulline will receive an initial intravenous bolus of 20 mg/kg (to a maximum of 1500 mg) L-citrulline over 10 minutes. The study solution will be prepared as a 5% isotonic solution (50 mg/mL) in 5% dextrose water. Immediately after the initial bolus, a continuous intravenous infusion of L-citrulline at 9 mg/kg (max 700 mg) per hour will be administered through a dedicated intravenous line or port of a multi-lumen catheter.
  Interventions: Drug: L-Citrulline
- Placebo Arm (Placebo Comparator): Patients randomized to placebo arm will receive an infusion of 5% dextrose water matched for volume and color to the citrulline infusion. The placebo infusion will consist of an initial iv bolus (up to 30 mL) over 10 minutes followed by a continuous infusion of 5% dextrose water (about 15 mL/hr). The initial bolus and subsequent infusion will be administered through a dedicated intravenous line or port of a multi-lumen catheter.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: L-Citrulline — L-Citrulline (Turnobi) for Injection. Patients will receive an initial bolus of 20 mg/kg (maximum 1500 mg), followed by study infusion of 9 mg/kg per hour (maximum 700mg) for up to 10 days.
  Other Names: L-CIT, CIT
  Arms: IV L-Citrulline (Turnobi) Arm
Drug: Placebo — Patients randomized to placebo will receive equal volume bolus and study infusion of 5% dextrose water for a maximum of 10 days.
  Arms: Placebo Arm

SUMMARY:
Prospective, Randomized, Double-Blind, Placebo-Controlled Phase II Trial of Intravenous L-Citrulline (Turnobi) to Delay and Potentially Prevent the Need for Invasive Mechanical Ventilation for Acute Hypoxemic Respiratory Failure in Patients with COVID-19 (SARS-CoV2) Illness. To evaluate safety and efficacy of a bolus loading dose and continuous intravenous infusion of L-Citrulline compared to placebo in patients hospitalized with COVID-19 infection (SARS-CoV-2).

DETAILED DESCRIPTION:
Intravenous L-citrulline (Turnobi) administration will safely restore the homeostasis of nitric oxide synthase by increasing both plasma citrulline and arginine levels. Investigators also reason that restoration of citrulline/arginine balance through citrulline administration will safely re-establish homeostasis of NOS, lower oxidative stress, and reduce inflammation, thereby delaying and potentially preventing the need for invasive mechanical ventilation in participants hospitalized with COVID-19 infection (SARS-CoV-2). The body lives in a delicate balance of homeostasis. The urea/NO cycle plays a critical role in maintaining redox homeostasis and as such, also plays a role in regulating inflammation. The biochemical relationships are complex and depend on inter-organ transfer, membrane transport, and intracellular compartmentation. However, data above demonstrate that citrulline, arginine, and NO are critical in maintaining this homeostasis through their regulation of NOS. Inflammation, especially from infection, results in decreased activity of CPS1 and increased activity of arginase, which decreases levels of both citrulline and arginine. These decreased levels result in dysregulated and uncoupled NOS, which drives both overexuberant NO production and formation of ROS. Both the NO production and ROS further exacerbate the inflammatory cascade, resulting in other organ dysfunctions, including acute lung injury. Both inflammation and oxidative stress have been shown to be driving forces for the development of ALI and regulated NOS function is vital to reducing both. Both plasma citrulline and arginine are deficient in sepsis and levels are inversely associated with development of ALI. Furthermore, citrulline replacement safely increases plasma levels of both citrulline and arginine in healthy volunteers, BMT patients, adults with sepsis, children with sickle cell disease, and children after congenital heart surgery. It seems highly likely that citrulline therapy in the setting of COVID-19 (SARS-CoV2) induced acute hypoxemic respiratory illness will safely increase citrulline and arginine levels and help re-establish NOS homeostasis, resulting in NO production in compartments that are more homeostatically appropriate so as to reduce pulmonary vascular resistance and enhance coupling of NOS to minimize superoxide production thus reducing free radical mediated ALI.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years.
2. Clinical evidence of COVID-19 (SARS-CoV2) infection, defined as a positive COVID-19 laboratory test plus evidence of an acute hypoxemic respiratory illness requiring oxygen.
3. Admitted and transferred to floor without intubation.

Exclusion Criteria:

1. No consent/inability to obtain consent
2. Patient, surrogate, or physician not committed to full support
3. Malignant or other irreversible condition and estimated 28-day mortality ≥ 50%
4. Moribund patient not expected to survive 48 hours (as defined by primary medical team) from start of study infusion
5. End-stage Liver Disease as defined by Child-Pugh Score > 9
6. Currently enrolled in, or participated in another study of an investigational compound within the last 30 days
7. Pregnant female, or female who is breast feeding
8. Allergy to L-citrulline or arginine or any citrulline- or arginine-containing product
9. Patient not otherwise suitable for the study in the opinion of any of the investigators
10. Requirement for intubation and invasive mechanical ventilation before study enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gurdyal Kalsi, MD, MFPM, Study Director — Asklepion Pharmaceuticals, LLC
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IV L-Citrulline (Turnobi) Arm | Placebo Arm
Started | 33 | 32
Completed | 22 | 23
Not Completed | 11 | 9
Not completed — Adverse Event | 2 | 1
Not completed — Death | 2 | 5
Not completed — Lost to Follow-up | 1 | 0
Not completed — Other | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Sponsor Decision | 1 | 0
Not completed — Withdrawal by Subject | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IV L-Citrulline (Turnobi) Arm | Placebo Arm | Total
Number analyzed (Participants) | 33 | 32 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.30 (11.04) | 51.13 (10.34) | 50.71 (10.63)
Age, Customized [Count of Participants; unit: Participants]
  18-49 years | 13 | 12 | 25
  50-65 years | 20 | 20 | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 9 | 25
  Male | 17 | 23 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 29 | 26 | 55
  Unknown or Not Reported | 1 | 4 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 17 | 35
  White | 12 | 12 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Time to Non-invasive/Invasive Mechanical Ventilation
Description: Time in hours from the initiation of the treatment until mechanical ventilation is required, whether non-invasive (e.g., high flow nasal cannula, bilevel positive airway pressure, oxygen therapy) or invasive (i.e., requiring intubation).
Time Frame: From the start of infusion to Day 60 Follow-up
Population: Patients in the Intent-to-treat population that required invasive or non-invasive ventilation.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | IV L-Citrulline (Turnobi) Arm | Placebo Arm
Number analyzed (Participants) | 11 | 10
Hours | 96.65 (143.73) | 70.49 (62.44)
Statistical Analysis 1: Comparison: IV L-Citrulline (Turnobi) Arm vs Placebo Arm; Test type: Other; p = 0.782, Log Rank; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.45 to 2.86]
Statistical Analysis 2: Comparison: IV L-Citrulline (Turnobi) Arm vs Placebo Arm; Test type: Other; p = 0.668, Regression, Logistic; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.46 to 3.40]

2. Primary Outcome: Time to Non-invasive Mechanical Ventilation
Description: Time in hours from the initiation of the treatment until non-invasive mechanical ventilation is required (e.g., high flow nasal cannula, bilevel positive airway pressure, oxygen therapy) .
Time Frame: From the start of infusion to Day 60 Follow-up
Population: Patients in the Intent-to-treat population requiring non-invasive mechanical ventilation.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | IV L-Citrulline (Turnobi) Arm | Placebo Arm
Number analyzed (Participants) | 9 | 8
Hours | 66.17 (105.40) | 105.70 (108.90)
Statistical Analysis 1: Comparison: IV L-Citrulline (Turnobi) Arm vs Placebo Arm; Test type: Other; p = 0.360, Log Rank; Hazard Ratio (HR) = 1.58, 95% CI 2-sided [0.59 to 4.22]

3. Primary Outcome: Time to Invasive Mechanical Ventilation
Description: Time in hours from the initiation of the treatment until intubation for invasive mechanical ventilation is required.
Time Frame: From the start of infusion to Day 60 Follow-up
Population: Patients in the Intent-to-treat population requiring intubation for invasive mechanical ventilation.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | IV L-Citrulline (Turnobi) Arm | Placebo Arm
Number analyzed (Participants) | 4 | 6
Hours | 290.01 (254.31) | 148.07 (108.08)
Statistical Analysis 1: Comparison: IV L-Citrulline (Turnobi) Arm vs Placebo Arm; Test type: Other; p = 0.285, Log Rank; Hazard Ratio (HR) = 0.49, 95% CI 2-sided [0.13 to 1.83]
Statistical Analysis 2: Comparison: IV L-Citrulline (Turnobi) Arm vs Placebo Arm; Test type: Other; p = 0.471, Regression, Logistic; Odds Ratio (OR) = 0.60, 95% CI 2-sided [0.15 to 2.41]

4. Primary Outcome: Systolic Blood Pressure
Description: Systolic blood pressure measured in mmHg
Time Frame: Day 1
Population: Patients in the safety population with measurement(s) of systolic blood pressure
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | IV L-Citrulline (Turnobi) Arm | Placebo Arm
Number analyzed (Participants) | 24 | 27
Millimeters of mercury | 118.63 (14.69) | 130.19 (15.71)

5. Primary Outcome: Diastolic Blood Pressure
Description: Diastolic blood pressure measured in mmHg
Time Frame: Day 1
Population: Patients in the safety population with measurement(s) of diastolic blood pressure
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | IV L-Citrulline (Turnobi) Arm | Placebo Arm
Number analyzed (Participants) | 24 | 27
Millimeters of mercury | 73.58 (10.06) | 79.74 (13.13)

6. Primary Outcome: Mean Arterial Pressure
Description: Mean arterial pressure measured in mmHg
Time Frame: Day 1
Population: Patients in the safety population with measurement(s) of mean arterial blood pressure
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | IV L-Citrulline (Turnobi) Arm | Placebo Arm
Number analyzed (Participants) | 24 | 27
Millimeters of mercury | 87.58 (10.03) | 94.30 (13.49)

7. Secondary Outcome: Blood Levels of Arginine
Description: Plasma levels of arginine
Time Frame: Plasma levels of arginine at 0, 2 and 12 hours, and 2, 4, 6, 8, 10 days after initiation of treatment
Population: Patients with at least 1 measurement of plasma arginine
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | IV L-Citrulline (Turnobi) Arm | Placebo Arm
Number analyzed (Participants) | 33 | 32
µmol/L
  Hour 0: number analyzed (Participants) | 30 | 30
  Hour 0 | 67.6 (28.27) | 67.88 (29.51)
  Hour 2: number analyzed (Participants) | 30 | 30
  Hour 2 | 92.57 (30.84) | 71.51 (29.15)
  Hour 12: number analyzed (Participants) | 29 | 29
  Hour 12 | 128.11 (41.3) | 75.7 (24.54)
  Day 2: number analyzed (Participants) | 23 | 27
  Day 2 | 142.02 (54.51) | 82.19 (26.33)
  Day 4: number analyzed (Participants) | 14 | 20
  Day 4 | 152.00 (66.7) | 79.66 (22.84)
  Day 6: number analyzed (Participants) | 7 | 12
  Day 6 | 169.33 (113.62) | 70.78 (19.46)
  Day 8: number analyzed (Participants) | 10 | 9
  Day 8 | 167.64 (82.5) | 81.79 (32.28)
  Day 10: number analyzed (Participants) | 9 | 7
  Day 10 | 160.02 (83.39) | 83.9 (37.36)

8. Secondary Outcome: Blood Levels of Citrulline
Description: Plasma levels of citrulline
Time Frame: Plasma levels of citrulline at 0, 2 and 12 hours, and 2, 4, 6, 8, 10 days after initiation of treatment
Population: All patients with at least 1 plasma citrulline measurement
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | IV L-Citrulline (Turnobi) Arm | Placebo Arm
Number analyzed (Participants) | 33 | 32
µmol/L
  Hour 0: number analyzed (Participants) | 30 | 30
  Hour 0 | 24.64 (25.91) | 18.08 (13.7)
  Hour 2: number analyzed (Participants) | 30 | 30
  Hour 2 | 1094.41 (2463.97) | 18.39 (14.08)
  Hour 12: number analyzed (Participants) | 29 | 29
  Hour 12 | 997.61 (2133.07) | 21.84 (16.14)
  Day 2: number analyzed (Participants) | 23 | 27
  Day 2 | 278.2 (353.32) | 24.68 (27.57)
  Day 4: number analyzed (Participants) | 14 | 20
  Day 4 | 626.33 (1562.95) | 20.53 (15.84)
  Day 6: number analyzed (Participants) | 7 | 12
  Day 6 | 185.14 (68.63) | 20.96 (10.16)
  Day 8: number analyzed (Participants) | 10 | 9
  Day 8 | 192.72 (127.72) | 24.84 (9.64)
  Day 10: number analyzed (Participants) | 9 | 7
  Day 10 | 206.26 (135.94) | 24.56 (11.46)

9. Secondary Outcome: Evaluate the Effect of Intravenous L-Citrulline Compared to Placebo as Measured by the Total Length of All Mechanical Ventilation
Description: Total length of time of any mechanical ventilation
Time Frame: Day 1 through Day 60 Follow Up
Population: Patients in the Intent-to-treat population requiring mechanical ventilation
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | IV L-Citrulline (Turnobi) Arm | Placebo Arm
Number analyzed (Participants) | 14 | 12
Hours | 270.91 (304.03) | 451.87 (503.68)
Statistical Analysis 1: Comparison: IV L-Citrulline (Turnobi) Arm vs Placebo Arm; Test type: Other; p = 0.668, Zero-inflated negative binomial analyses; Odds Ratio, log = 0.81, 95% CI 2-sided [0.30 to 2.20]
Statistical Analysis 2: Comparison: IV L-Citrulline (Turnobi) Arm vs Placebo Arm; Test type: Other; p = 0.437, Zero-inflated negative binomial analyses; Incidence Rate Ratio = 0.66, 95% CI 2-sided [0.23 to 1.90]

10. Secondary Outcome: Evaluate the Effect of IV L-Citrulline to Placebo for Hospital All Cause Mortality
Description: To evaluate the effect of intravenous L-Citrulline compared to placebo on Hospital all-cause mortality
Time Frame: Day 1 through day 12
Population: Intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | IV L-Citrulline (Turnobi) Arm | Placebo Arm
Number analyzed (Participants) | 33 | 32
Participants | 2 | 5
Statistical Analysis 1: Comparison: IV L-Citrulline (Turnobi) Arm vs Placebo Arm; Test type: Other; p = 0.232, Regression, Logistic; Odds Ratio (OR) = 0.35, 95% CI 2-sided [0.06 to 1.97]

11. Secondary Outcome: Percentage of Patients Admitted to Intensive Care
Time Frame: Day 1 through Day 12 (DC)
Population: Intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | IV L-Citrulline (Turnobi) Arm | Placebo Arm
Number analyzed (Participants) | 33 | 32
Participants | 12 | 13
Statistical Analysis 1: Comparison: IV L-Citrulline (Turnobi) Arm vs Placebo Arm; Test type: Other; p = 0.729, Regression, Logistic; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.31 to 2.28]

12. Secondary Outcome: Duration of Intensive Care Unit (ICU) Stay
Description: Length of ICU stay (days)
Time Frame: From admission to ICU until discharge or death
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | IV L-Citrulline (Turnobi) Arm | Placebo Arm
Number analyzed (Participants) | 12 | 13
Days | 14.83 (12.29) | 17.31 (18.87)
Statistical Analysis 1: Comparison: IV L-Citrulline (Turnobi) Arm vs Placebo Arm; Test type: Other; p = 0.706, Zero-inflated negative binomial analyses; Odds Ratio, log = 1.22, 95% CI 2-sided [0.43 to 3.44]
Statistical Analysis 2: Comparison: IV L-Citrulline (Turnobi) Arm vs Placebo Arm; Test type: Other; p = 0.788, Zero-inflated negative binomial analyses; Incidence Rate Ratio = 1.12, 95% CI 2-sided [0.49 to 2.56]

13. Secondary Outcome: Duration of Hospitalisation
Description: Length of hospital stay (days)
Time Frame: From admission to hospital until discharge or death
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | IV L-Citrulline (Turnobi) Arm | Placebo Arm
Number analyzed (Participants) | 33 | 32
Days | 10.61 (12.74) | 11.88 (14.29)
Statistical Analysis 1: Comparison: IV L-Citrulline (Turnobi) Arm vs Placebo Arm; Test type: Other; p = 0.834, Negative binomial analysis; Incidence Rate Ratio = 1.08, 95% CI 2-sided [0.52 to 2.25]

14. Secondary Outcome: Number of Patients Requiring Intubation
Description: Percentage of patients requiring any mechanical ventilation, invasive mechanical ventilation and non-invasive mechanical ventilation.
Time Frame: From the start of infusion to Day 60 Follow-up
Population: Intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | IV L-Citrulline (Turnobi) Arm | Placebo Arm
Number analyzed (Participants) | 33 | 32
Participants
  Non-invasive/invasive mechanical ventilation | 14 | 12
  Non-invasive mechanical ventilation | 12 | 10
  Invasive mechanical ventilation | 4 | 6

15. Secondary Outcome: Overall Duration of Mechanical Ventilation
Description: Total time on any mechanical ventilation, invasive mechanical ventilation, non-invasive mechanical ventilation and nasal cannula
Time Frame: From the start of infusion to Day 60 Follow-up
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | IV L-Citrulline (Turnobi) Arm | Placebo Arm
Number analyzed (Participants) | 33 | 32
Hours
  Total time on mechanical ventilation: number analyzed (Participants) | 14 | 12
  Total time on mechanical ventilation | 239.31 (243.08) | 222.08 (370.90)
  Total time of non-invasive mechanical ventilation: number analyzed (Participants) | 12 | 10
  Total time of non-invasive mechanical ventilation | 224.64 (254.22) | 219.27 (309.40)
  Total time of invasive mechanical ventilation: number analyzed (Participants) | 4 | 6
  Total time of invasive mechanical ventilation | 274.27 (158.86) | 538.28 (469.21)
  Total time on Nasal Cannula: number analyzed (Participants) | 9 | 7
  Total time on Nasal Cannula | 239.31 (243.08) | 222.08 (370.90)

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the time that the participant was first administered the study infusion (study hour = 0) until Day 10. Adverse events spontaneously reported to the investigator or observed by the investigator after Day 10 until Day 60 Follow Up were also collected and recorded.
Description: All available clinical data were monitored for AEs. Clinically important/unexpected adverse experiences were recorded as AEs.
  Clinical outcomes of acute hypoxemic respiratory illness progressing to critical illness due to COVID-19 were not considered AEs and therefore not collected or reported.
  A Vasopressor Dependency Index was calculated at baseline, 60 minutes after completion of the bolus, and every 4 hours during infusion. An increase in VDI of >33% from baseline was considered as an AE.
Arm/Group | IV L-Citrulline (Turnobi) Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 2/33 | 5/32
Serious Adverse Events (participants affected / at risk) | 6/33 | 10/32
Other Adverse Events (participants affected / at risk) | 11/33 | 11/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IV L-Citrulline (Turnobi) Arm (N=33) | Placebo Arm (N=32)
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Cardiac failure; metabolic acidosis (Cardiac disorders) | 1 | 0
Chest pain; Dyspnoea; COVID-19 (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Intracranial hemorrhage (Vascular disorders) | 1 | 1
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0
Status epilepticus (Nervous system disorders) | 1 | 0
Syncope (Cardiac disorders) | 1 | 0
Acute Respiratory Distress Syndrome, Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute kidney injury; renal tubular necrosis (Renal and urinary disorders) | 0 | 1
Brain Injury (Nervous system disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 2
Cardiac valve vegetation (Cardiac disorders) | 0 | 1
Cardio-respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV L-Citrulline (Turnobi) Arm (N=33) | Placebo Arm (N=32)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2)
Chest Pain (General disorders) | 0 (0) | 1 (1)
Clostridium Difficile Infection (Infections and infestations) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 2 (2) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Endocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Enterococcal Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal Infection (Infections and infestations) | 1 (1) | 1 (1)
Enterococcus Test Positive (Investigations) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Infusion Site Reaction (General disorders) | 3 (3) | 2 (2)
Ischaemic Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Lactic Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Liver Function Test Increased (Investigations) | 0 (0) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Skin Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Staphylococcal Sepsis; Alpha Haemolytic Streptococcal Infection (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous Emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Troponin I Increased (Investigations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 0 (0)
Ventricular Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-06-15): https://cdn.clinicaltrials.gov/large-docs/84/NCT04570384/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-16): https://cdn.clinicaltrials.gov/large-docs/84/NCT04570384/SAP_001.pdf